CLINICAL TRIAL: NCT07016373
Title: Effect of Topical Application of Medical Grade Manuka Honey on Pain Intensity and Tissue Healing After Palatal Epithelial-connective Tissue Graft Harvesting: a Double-blinded Randomised Controlled Trial
Brief Title: Role of Manuka Honey in Lowering Pain and Boosting Healing After Gum Graft Surgery.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Mouradian (Other)
Responsible Party: Sponsor-Investigator, Nancy Mouradian, Clinical Professor, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-471 / 28-11-2024
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Gingival Recession, Mucogingival Surgery
Keywords: mucogingival surgery; recession; gingival graft; palatal donor site; medical grade manuka honey; healing; pain
MeSH Terms: conditions — Gingival Recession; Pain

STUDY DESIGN:
Intervention Model Description: This is a split-mouth model where the patient will be their own control, receiving two surgeries but with different post-operative care.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery A with Honey/ Surgery B without Honey (Experimental): Surgeries A and B will be performed 4 weeks apart. During both surgeries, recipient sites will be distant from donor sites (mandibular recipient site and palatal donor site). A safety distance of 2 mm from the marginal gingiva should be maintained during incisions. Glandular and fatty tissue will be removed from the graft, which may or may not be de-epithelialized depending on the procedure for which it was harvested. It will then be adapted to the recipient site and sutured in place. During post-operative healing, surgery A will include a palatal plate with Manuka honey . Surgery B will include a palatal plate without Manuka Honey.
  Interventions: Device: Palatal Plate without Manuka Honey; Device: Palatal plate with Manuka Honey
- Surgery A without Honey/ Surgery B with Honey (Experimental): Surgeries A and B will be performed 4 weeks apart. During both surgeries, recipient sites will be distant from donor sites (mandibular recipient site and palatal donor site). A safety distance of 2 mm from the marginal gingiva should be maintained during incisions. Glandular and fatty tissue will be removed from the graft, which may or may not be de-epithelialized depending on the procedure for which it was harvested. It will then be adapted to the recipient site and sutured in place. During post-operative healing, surgery A will include a palatal plate without Manuka honey . Surgery B will include a palatal plate with Manuka Honey.
  Interventions: Device: Palatal Plate without Manuka Honey; Device: Palatal plate with Manuka Honey

INTERVENTIONS:
Device: Palatal Plate without Manuka Honey — A Palatal plate without Manuka Honey will be inserted by a blinded investigator on the donor site for post-operative procedures.
Device: Palatal plate with Manuka Honey — A Palatal plate with Manuka Honey will be inserted by a blinded researcher on the donor site.

SUMMARY:
The goal of this clinical trial is to learn if medical grade Manuka Honey works to lower pain and improve healing sites after gum grafting surgery. The main questions are:

* Does medical grade Manuka honey lower pain and painkiller use after gum grafting surgery ?
* Does medical grade Manuka honey boost healing after gum grafting surgery ?

Researchers will compare, within the same patient, the results of a surgery with the application of Manuka honey in a retainer to a surgery without the application of honey in the retainer for the healing period.

Participants will:

* Visit the clinic for their first surgery.
* Fill up a daily survey to explain their level of pain and the amount of painkiller drugs used.
* Visit the clinic once every week for 6 weeks for follow-ups.
* Visit the clinic for their second surgery, four weeks after the first one.
* Fill up a daily survey to explain their level of pain and the amount of painkiller drugs used after the second surgery.
* Visit the clinic once every week for 6 weeks for follow-ups on the second surgery
* Fill a survey to compare both surgeries .
* Visit the clinic 2 months, 6 months and one year after the surgeries for more follow-ups.

DETAILED DESCRIPTION:
The study aims to identify if medical grade Manuka honey applied to the donor site has an impact on:

* postoperative pain using a visual analogue scale and by assessing patients' consumption of analgesics
* wound healing using the Landry Wound Healing Index and the hydrogen peroxide test which detects the level of epithelialisation of the wound (incomplete or complete).

During the preoperative phase, an initial periodontal assessment will be made to determine the eligibility of patients to participate in the study according to the inclusion and exclusion criteria. Depending on their needs, the 24 participants will receive supra and/or sub-gingival scaling at least four weeks prior to the first surgery. An alginate impression of the maxilla will be taken for all participants for the fabrication of the palatal plate.

Immediately prior to surgery, participants will gargle with a 0.12% chlorhexidine gluconate mouthwash for one minute and will receive a 600 mg ibuprofen tablet . They will be instructed to take another 600 mg ibuprofen tablet six hours later. Participants will receive two surgeries with a palatal harvest (one on each side of the palate). The recipient site will be prepared conventionally. During surgery, recipient sites will be distant from donor sites (mandibular recipient site and palatal donor site). A safety distance of 2 mm from the marginal gingiva should be maintained during incisions. Glandular and fatty tissue will be removed from the graft, which may or may not be de-epithelialized depending on the procedure for which it was harvested. It will then be adapted to the recipient site and sutured in place. The dimensions of the graft and of the wound at the donor site will be measured using a UNC 15 probe. Primary contraction can then be assessed. The residual thickness of the palatal tissue will also be assessed at this time, using a 30C anaesthetic needle, to which we will add a rubber stopper for an endodontic file. Measurement is then taken using an endodontic ruler.

For the healing period of one of the gingival grafts, the patient will wear a palatal plate with medical grade Manuka honey, and, for the other gingival graft, the patient will wear a palatal plate without a topical agent. A refractory period of at least four weeks will be observed between procedures. The palatal plate will be maintained for 7 days. A different clinician will insert and remove the palatal plate to preserve double blinding.

The usual post-operative instructions for mucogingival surgery will be given verbally and in leaflet form to the participant. A prescription for ibuprofen and chlorhexidine gluconate 0.12% mouthwash will be given to the patient.

Participants will be required to complete the roadmap provided for 14 days following each intervention. Clinical follow-ups will take place at 1, 2, 3, 4 and 6 weeks and at 2, 6 and 12 months post-operatively. We will also measure the dimensions of the palatal wound at these follow-ups. At 2, 6 and 12 months, we will measure the width of keratinised tissue and root coverage obtained.

ELIGIBILITY:
Inclusion Criteria:

Participants must :

* Be 18 years of age or older.
* Be in good systemic health or have well-controlled systemic health.
* Have a healthy or stable periodontium after conventional periodontal treatment.
* Have good clinical gingival health or gingivitis on an intact or reduced periodontium, with or without a history of periodontitis
* Maintain good oral hygiene.
* Have a simplified plaque index and gingival bleeding index below 20%
* Require two mucogingival surgeries involving bilateral epithelial-conjunctival graft harvesting (free gingival graft or de-epithelialised connective tissue graft).
* The surgeries must treat single or multiple gingival recessions, or mucogingival defects around teeth or implants.

Exclusion Criteria:

* Smokers or users of other tobacco products
* Pregnant participants
* Participants who are uncooperative or have a psychological condition that makes free and informed consent or compliance with instructions impossible
* Participants with a condition that impairs healing (e.g. poorly controlled diabetes, coagulation disorder, etc.) or the objective assessment of pain at the sampling site (e.g. autoimmune diseases, orofacial pain, etc.)
* Participants regularly taking the following medications : non-steroidal anti-inflammatory drugs, bisphosphonates, sedatives, psychotropic drugs and corticosteroids.
* During the study, those who develop a condition that interferes with healing, become smokers, start medication that acts on the central nervous system, do not adhere strictly to instructions or do not respect follow-ups.
* Participants who have already received a palatal surgery in the past or whose palatal tissue thickness is less than 3 mm will not be excluded, to allow comparative analyses in sub-groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-12-26 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient Pain Level | Pain levels will be assessed daily for 14 days
  Patient's percieved pain levels will be measured daily at the exact same hour for 14 days with a survey, where they will indicate:
  Their pain levels with a visual analog scale ranging from 0 to 10. 0 indicates no pain and 10 indicates the maximum pain imaginable.
Daily Ibuprofen Intake | Pain levels will be assessed daily for 14 days
  Patient's ibuprofen intake will be declared daily at the exact same hour for 14 days with a survey, where they will indicate The daily intake of ibuprofen tablets (n of tablets taken during the day)

SECONDARY OUTCOMES:
Landry Wound Index | It will be determined at 1, 2, 3, 4, 6 weeks, 2 months.
  Palatal wound healing will be evaluated by the clinician himself using the Landry Wound Healing Index, an index that tests healing with specific criteria like tissue color, palpation response, incision margin and the extent of the wound. This index is a scale from 1 to 5 where 1 is very poor healing and 5 is excellent healing.
Bubbling Test | It will be measured at 1, 2, 3, 4, 6 weeks, 2 months.
  Palatal wound healing will also be evaluated by the clinician himself using the Bubbling test that uses hydrogen peroxide at 3% to determine if the tissue re-epithelialized completely. The presence of bubbles indicates that the wound did not epithelialize completely yet. Absence of bubbles indicates complete epithelialization. This will be measured dichotomously with 0 being incomplete epithelialization and 1 being complete epithelialization.
Keratinized tissue width | ,Keratinized tissue width will be measured at 2, 6 and 12 months.
  Keratinized tissue width (in mm) and will be assessed at 2, 6 and 12 months. It is typically measured from the gingival margin to the mucogingival junction using a periodontal probe.
Root Coverage | Root coverage will be measured at 2, 6 and 12 months
  Root coverage (in %) will be assessed at 2, 6 and 12 months. We will initially measure the depth of recession (in mm), and will do so at the designated time frames. The difference between initial and follow-up measures will then be reported as a percentage of the initial measurement.
Other complications | Other complications will be assessed daily for 14 days
  The other complications will be part of the pain level survey that will be filled by patients, where they will indicate if they feel any other sort of complications. It will be a qualitative outcome to bring more accuracy to patients' experience with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mouradian, DMD, MSc, FRCD(C), Dip.ABP, Study Director — Laval University; Benjamin Labelle, DMD, MSc, Cert. Perio, FRCD(C), Study Director
Locations (1):
- Laval university- Faculty of Dentistry, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tavelli L, Asa'ad F, Acunzo R, Pagni G, Consonni D, Rasperini G. Minimizing Patient Morbidity Following Palatal Gingival Harvesting: A Randomized Controlled Clinical Study. Int J Periodontics Restorative Dent. 2018 Nov/Dec;38(6):e127-e134. doi: 10.11607/prd.3581. PMID 30304077
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Background] Rajapakse PS, McCracken GI, Gwynnett E, Steen ND, Guentsch A, Heasman PA. Does tooth brushing influence the development and progression of non-inflammatory gingival recession? A systematic review. J Clin Periodontol. 2007 Dec;34(12):1046-61. doi: 10.1111/j.1600-051X.2007.01149.x. Epub 2007 Oct 22. PMID 17953693
- [Background] Lost C. Depth of alveolar bone dehiscences in relation to gingival recessions. J Clin Periodontol. 1984 Oct;11(9):583-9. doi: 10.1111/j.1600-051x.1984.tb00911.x. PMID 6593330
- [Background] Serino G, Wennstrom JL, Lindhe J, Eneroth L. The prevalence and distribution of gingival recession in subjects with a high standard of oral hygiene. J Clin Periodontol. 1994 Jan;21(1):57-63. doi: 10.1111/j.1600-051x.1994.tb00278.x. PMID 8126246
- [Background] Kennedy JE, Bird WC, Palcanis KG, Dorfman HS. A longitudinal evaluation of varying widths of attached gingiva. J Clin Periodontol. 1985 Sep;12(8):667-75. doi: 10.1111/j.1600-051x.1985.tb00938.x. PMID 3902907
- [Background] Wennstrom JL. Lack of association between width of attached gingiva and development of soft tissue recession. A 5-year longitudinal study. J Clin Periodontol. 1987 Mar;14(3):181-4. doi: 10.1111/j.1600-051x.1987.tb00964.x. PMID 3470324
- [Background] Cortellini P, Bissada NF. Mucogingival conditions in the natural dentition: Narrative review, case definitions, and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S204-S213. doi: 10.1002/JPER.16-0671. PMID 29926948
- [Background] Chambrone L, Tatakis DN. Long-Term Outcomes of Untreated Buccal Gingival Recessions: A Systematic Review and Meta-Analysis. J Periodontol. 2016 Jul;87(7):796-808. doi: 10.1902/jop.2016.150625. Epub 2016 Feb 15. PMID 26878749
- [Background] Romandini M, Soldini MC, Montero E, Sanz M. Epidemiology of mid-buccal gingival recessions in NHANES according to the 2018 World Workshop Classification System. J Clin Periodontol. 2020 Oct;47(10):1180-1190. doi: 10.1111/jcpe.13353. Epub 2020 Sep 2. PMID 32748539
- [Background] Kassab MM, Cohen RE. The etiology and prevalence of gingival recession. J Am Dent Assoc. 2003 Feb;134(2):220-5. doi: 10.14219/jada.archive.2003.0137. PMID 12636127
- [Background] Albandar JM, Kingman A. Gingival recession, gingival bleeding, and dental calculus in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):30-43. doi: 10.1902/jop.1999.70.1.30. PMID 10052768
- [Background] Lava-Sanchez PA, Puppo S. Occurrence in vivo of "hidden breaks" at specific sites of 26 S ribosomal RNA of Musca carnaria. J Mol Biol. 1975 Jun 15;95(1):9-20. doi: 10.1016/0022-2836(75)90331-9. No abstract available. PMID 1152058
- [Background] Agossa K, Godel G, Dubar M, S Y K, Behin P, Delcourt-Debruyne E. Does Evidence Support a Combined Restorative Surgical Approach for the Treatment of Gingival Recessions Associated With Noncarious Cervical Lesions? J Evid Based Dent Pract. 2017 Sep;17(3):226-238. doi: 10.1016/j.jebdp.2017.04.001. Epub 2017 Apr 11. PMID 28865819
- [Background] Yupanqui Mieles J, Vyas C, Aslan E, Humphreys G, Diver C, Bartolo P. Honey: An Advanced Antimicrobial and Wound Healing Biomaterial for Tissue Engineering Applications. Pharmaceutics. 2022 Aug 10;14(8):1663. doi: 10.3390/pharmaceutics14081663. PMID 36015289
- [Background] Tavelli L, Barootchi S, Stefanini M, Zucchelli G, Giannobile WV, Wang HL. Wound healing dynamics, morbidity, and complications of palatal soft-tissue harvesting. Periodontol 2000. 2023 Jun;92(1):90-119. doi: 10.1111/prd.12466. Epub 2022 Dec 30. PMID 36583690
- [Background] Carter DA, Blair SE, Cokcetin NN, Bouzo D, Brooks P, Schothauer R, Harry EJ. Therapeutic Manuka Honey: No Longer So Alternative. Front Microbiol. 2016 Apr 20;7:569. doi: 10.3389/fmicb.2016.00569. eCollection 2016. PMID 27148246
- [Background] Alasqah M, Alrashidi A, Alshammari N, Alshehri A, Gufran K. Effect of honey dressing material on palatal wound healing after harvesting a free gingival graft: a prospective randomized case control study. Eur Rev Med Pharmacol Sci. 2022 Apr;26(8):2662-2668. doi: 10.26355/eurrev_202204_28595. PMID 35503610